CLINICAL TRIAL: NCT01039857
Title: Does an Integrative Neuro-psychotherapy Program Foster the Adjustment in Depressed Stroke Patients? A Randomized Controlled Study.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Project end after 3 years; prolongation was rejected
Sponsor: University of Bern (Other)
Collaborators: Swiss National Science Foundation (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Prof. Dr. Hansjoerg Znoj, University of Bern, Department of Clinical Psychology and Psychotherapy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012/08; 100014-124574, 2009-2012 (Other Grant/Funding Number: SNF); 1784 (Other: Bern University Hospital)
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Adjustment Disorders; Non-progressive Brain Injury
Keywords: Psychotherapy; Depression; Adjustment Disorders; Neuropsychology; Rehabilitation; Coping Skills; Stroke; Caregivers
MeSH Terms: conditions — Adjustment Disorders; Depression; Stroke | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured solution focused therapy (Other): Neuropsychological Therapy, cognitive behavioral therapy, solution focused therapy
  Interventions: Behavioral: Neuropsychological Therapy, cognitive behavioral therapy, solution focused therapy
- Integrative clarification therapy (Experimental): Neuropsychological therapy, cognitive-behavioral therapy, emotion-focused techniques, clarification and interpersonal therapy techniques
  Interventions: Behavioral: Integrative Neuro-Psychotherapy

INTERVENTIONS:
Behavioral: Neuropsychological Therapy, cognitive behavioral therapy, solution focused therapy
  Arms: Structured solution focused therapy
Behavioral: Integrative Neuro-Psychotherapy — Neuropsychological therapy, cognitive-behavioral therapy, emotion-focused techniques, clarification and interpersonal therapy techniques
  Arms: Integrative clarification therapy

SUMMARY:
This is an intervention study with patients after a non-progressive brain injury who suffer from depression. It will determine whether an integration of neuropsychological and psychotherapeutic techniques and an additional caregivers support program offers benefits to those in the process of coping with the effects of a stroke. The investigators expect the integrative neuro-psychotherapy to be more effective in the treatment of emotional distress reactions following a stroke than the structured solution focused treatment.

DETAILED DESCRIPTION:
Background

A brain injury is one of the most common causes of disability acquired in adulthood. The full extent of the impairment usually only becomes clear during the course of rehabilitation. Apart from the emotional effects of dealing with the impairment, it is also invariably a matter of adjusting to life with a disability. In this phase of realization and coming to terms with their condition, many brain-injured people develop a mental disorder (mainly adjustment disorders with depressive and/or anxiety symptoms). Mental disorders related to adjustment are a significant and often limiting factor in patient rehabilitation. While there is a very extensive body of literature on the diagnosis and treatment of cognitive disorders following a brain injury, research on the diagnosis and treatment of clinical disorders following a brain injury is scarce. There are many theoretical observations in the available literature about ways of dealing with adjustment disorders following a brain injury in order to maximize a patient's rehabilitation outcome. Yet current research, based with randomized studies, is still in its infancy. The main aim of the current project is to close this scientific gap. A key objective of the proposed study is to investigate whether an integration of neuropsychological and psychotherapeutic techniques and an additional caregivers support program offers benefits to those in the process of coping with the effects of a brain injury.

It is expected that the integrative neuro-psychotherapy is more effective in the treatment of emotional distress reactions than the structured solution focused therapy. Moreover, a stronger improvement in acceptance, awareness, quality of life and goal attainment is anticipated in patients who receive the integrative neuro-psychotherapy treatment. A correlation is expected of the extent of improvement and neuropsychological functional level in memory and executive functioning. In addition, the extent of improvement might depend on personality changes due to the stroke or on the location and volume of the lesion.

Several measures will be used for patient assessment. Demographic data will be collected, MR or CT images will be made, the National Institute of Health Stroke Scale (NIHSS) will be applied. A comprehensive neuropsychological examination (memory, attention, executive functioning and visual functioning) will be performed with each patient before the beginning of the treatment. Several questionnaires measuring depressive symptoms, quality of life, coping strategies, awareness, personality changes, relationship and goals will be applied by patients, caregivers and therapists depending on the questionnaire.

Objective

A key objective of the proposed study is to investigate whether an integration of neuropsychological and psychotherapeutic techniques and an additional caregivers support program offers benefits to those in the process of coping with the effects of a non-progressive brain injury.

Methods

This is a randomized controlled intervention study with two treatment arms, the structured solution focused therapy and the integrative neuro-psychotherapy. 20 face to face sessions will be held for each patient. Primary caregivers will be supported by an online coaching tool. Assessments will be made at baseline, after 10 sessions (progress), after 20 sessions (termination) and at 6 months post treatment (follow-up). The hypothesis of statistically significant differences in the two groups will be tested by independent t-tests. Moreover, correlation tests will be applied to test post-hoc whether the extent of improvement measured by the BDI-II depends on the neuropsychological functional level in the cognitive area memory and executive functioning. A lesion analysis and estimation of the lesion volume will be carried out post-hoc in order to test whether these factors do predict the effectiveness of the integrative neuro-psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Non-progressive acquired brain injury
* Time passed since brain injury equal or more than 4 months
* Sufficient language ability to communicate and understand
* Sufficient language ability in German
* Currently in an outpatient setting
* Diagnosis of an adjustment disorder (DSM-IV: 309.x, acute or chronic)
* Age between 18 and 66 years

Exclusion Criteria

* Events other than non-progressive acquired brain injury (e.g. neurodegenerative illness)
* Presence of other chronic diseases (e.g. multiple sclerosis, sarcoidosis, Parkinson disorder, chronic pain disorder, rheumatic disorder)
* Moderate to severe cognitive impairment
* Prior history of psychiatric disease such as alcohol and drug abuse, personality disorders, obsessive-compulsive disorder, psychotic disorder
* Suicidal or violent behaviour

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
emotional distress measured by the Beck Depression Inventory (BDI-II) | after the first 10 sessions (Progress), end of therapy, 6 months after end of therapy (follow-up)

SECONDARY OUTCOMES:
Acceptance measured by the Trier Skala zur Krankheitsverarbeitung (TSK) | end of therapy, 6 months after end of therapy (follow-up)
Awareness measured by the Awareness Questionnaire | end of therapy, 6 months after end of therapy (follow-up)
Quality of life measured by the WHO Quality of Life-BREF (WHOQOL-BREF) | end of therapy, 6 months after end of therapy (follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Hansjoerg Znoj, Prof. Dr. phil., Study Chair — University of Bern, Dep. of Clinical Psychology and Psychotherapy; Helene Hofer, Dr. phil., Study Director — Bern University Hospital, Outpatient Clinic for Cognitive and Restorative Neurology; Martin Grosse Holtforth, Prof. Dr. phil., Study Director — University of Zurich, Dep. of Psychology, Research Unit Psychotherapy for Depression; Rene M Mueri, Prof. Dr. med., Study Director — Bern University Hospital, Outpatient Clinic for Cognitive and Restorative Neurology
Locations (1):
- Bern University Hospital Dep. for Cognitive and Restorative Neurology, Bern, Switzerland